CLINICAL TRIAL: NCT01149785
Title: A Phase 1, Fixed Sequence, Cross-Over Study To Estimate The Effect Of Multiple Doses Of Ketoconazole On The Single Dose Pharmacokinetics Of Crizotinib (PF-02341066) In Healthy Volunteers
Brief Title: Estimation Of Effect Of Ketoconazole On Pharmacokinetics Of Crizotinib In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: A8081015
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2011-10-19 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: crizotinib; healthy volunteers; ketoconazole; pharmacokinetics; single dose
MeSH Terms: interventions — Crizotinib; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): There should be at least 14-day washout period between treatment A and B.
  Interventions: Drug: crizotinib; Drug: ketoconazole

INTERVENTIONS:
Drug: crizotinib — Treatment A: a single 150-mg dose of crizotinib will be administered in the fasted state on Day 1 as 1 × 50-mg and 1 × 100-mg Immediate Release Tablets.
Drug: ketoconazole — Treatment B: 200 mg twice a day (approximately 12 hrs apart) doses of ketoconazole will be administered orally on an empty stomach from Day 1 to Day 16.
Drug: crizotinib — Treatment B: A single 150-mg dose of crizotinib will be administered in the fasted state on Day 4 as 1 × 50-mg and 1 × 100-mg Immediate Release Tablets.

SUMMARY:
The purpose of this study is to estimate the effect of multiple doses of ketoconazole on the single dose pharmacokinetics of crizotinib in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non-child bearing potential subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Subjects with evidence of disease, conditions affecting drug absorption, treatment with other investigational drug within 30 days, history of regular alcohol consumption, and use of prescription , nonprescription drugs and dietary supplement within 7 days, and blood donation of 500 mL within 56 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- [Derived] Xu H, O'Gorman M, Tan W, Brega N, Bello A. The effects of ketoconazole and rifampin on the single-dose pharmacokinetics of crizotinib in healthy subjects. Eur J Clin Pharmacol. 2015 Dec;71(12):1441-9. doi: 10.1007/s00228-015-1945-5. Epub 2015 Sep 18. PMID 26381275
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081015&StudyName=Estimation%20Of%20Effect%20Of%20Ketoconazole%20On%20Pharmacokinetics%20Of%20Crizotinib%20In%20Healthy%20Volunteers

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib 150 mg: Single oral dose of crizotinib 150 milligram (mg) immediate-release tablet (IRT) on Day 1 in first intervention period. A washout period of at least 14 days was maintained between each period.
- Crizotinib 150 mg + Ketoconazole 200 mg BID: Ketoconazole 200 mg tablet twice daily (BID), orally in fasted state from Day 1 to Day 16 and single oral dose of crizotinib 150 mg IRT on Day 4 in second intervention period. A washout period of at least 14 days was maintained between each period.
Period: First Intervention
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Started | 15 | 0
Completed | 15 | 0
Not Completed | 0 | 0
Period: Washout Period of at Least 14 Days
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Started | 15 | 0
Completed | 15 | 0
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Started | 0 | 15
Completed | 0 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive Crizotinib 150 mg IRT first and then Crizotinib 150 mg + Ketoconazole 200 mg BID
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 36.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)]
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0 (Pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hours (hrs) post crizotinib dose in period 1 and day 0, 0 (pre-dose), 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144, 192 and 312 hrs post crizotinib dose in period 2
Population: The pharmacokinetic (PK) parameter analysis population included all participants enrolled and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Crizotinib 150 mg: Single oral dose of crizotinib 150 mg IRT in first intervention period [Treatment A (Reference)].
- Crizotinib 150 mg + Ketoconazole 200 mg BID: Ketoconazole 200 mg tablet BID, orally in fasted state from Day 1 to Day 16 and single oral dose of crizotinib 150 mg IRT on Day 4 in second intervention period [Treatment B (Test)].
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
ng*hr/mL | 1260.00 (318.04) | 3986.00 (1010.10)
Statistical Analysis 1: Comparison: Crizotinib 150 mg vs Crizotinib 150 mg + Ketoconazole 200 mg BID; Natural log transformed AUC (0-∞) of crizotinib was analyzed using a mixed effect model with treatment as fixed effect and subject as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 316.36, 90% CI 2-sided [286.17 to 349.73]

2. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time Frame: 0 (Pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose in period 1 and day 0, 0 (pre-dose), 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144, 192 and 312 hrs post crizotinib dose in period 2
Population: The PK parameter analysis population included all participants enrolled and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
ng*hr/mL | 1197.00 (308.18) | 3929.00 (1004.40)
Statistical Analysis 1: Comparison: Crizotinib 150 mg vs Crizotinib 150 mg + Ketoconazole 200 mg BID; Natural log transformed AUClast of crizotinib was analyzed using a mixed effect model with treatment as fixed effect and subject as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 328.31, 90% CI 2-sided [296.42 to 363.63]

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
hr | 5.0 [2.0 to 5.0] | 6.0 [1.0 to 8.0]

4. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
hr | 37.1300 (4.3606) | 54.8700 (6.2589)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
ng/mL | 65.540 (24.486) | 94.470 (19.082)
Statistical Analysis 1: Comparison: Crizotinib 150 mg vs Crizotinib 150 mg + Ketoconazole 200 mg BID; Natural log transformed Cmax of crizotinib was analyzed using a mixed effect model with treatment as fixed effect and subject as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 144.13, 90% CI 2-sided [126.42 to 164.33]

6. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
L/hr | 122.600 (31.382) | 38.850 (10.413)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
L | 6580.0 (1881.8) | 3122.0 (1131.2)

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Crizotinib Metabolite (PF-06260182)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast) of crizotinib metabolite (PF-06260182).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
ng*hr/mL | 172.700 (56.751) | 897.400 (337.920)
Statistical Analysis 1: Comparison: Crizotinib 150 mg vs Crizotinib 150 mg + Ketoconazole 200 mg BID; Natural log transformed AUClast of crizotinib metabolite (PF-06260182) was analyzed using a mixed effect model with treatment as fixed effect and subject as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 519.65, 90% CI 2-sided [460.42 to 586.50]

9. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)] for Crizotinib Metabolite (PF-06260182)
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞) of crizotinib metabolite (PF-06260182).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
ng*hr/mL | 178.100 (57.989) | 920.600 (343.420)
Statistical Analysis 1: Comparison: Crizotinib 150 mg vs Crizotinib 150 mg + Ketoconazole 200 mg BID; Natural log transformed AUC (0-∞) of crizotinib metabolite (PF-06260182) was analyzed using a mixed effect model with treatment as fixed effect and subject as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 516.98, 90% CI 2-sided [457.88 to 583.72]

10. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
hr | 5.0 [4.0 to 6.0] | 8.0 [6.0 to 10.0]

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
ng/mL | 16.6900 (4.8538) | 26.9400 (5.4113)
Statistical Analysis 1: Comparison: Crizotinib 150 mg vs Crizotinib 150 mg + Ketoconazole 200 mg BID; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted Means = 161.42, 90% CI 2-sided [143.09 to 182.09]

12. Secondary Outcome: Metabolite to Parent Ratio of Area Under the Curve From Time Zero to Last Quantifiable Concentration for Crizotinib Metabolite Ratio (MRAUClast)
Description: Molar ratio of metabolite to parent area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (MRAUClast).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
Ratio | 0.1399 (0.0194) | 0.2217 (0.0397)

13. Secondary Outcome: Metabolite to Parent Ratio of Area Under the Curve From Time Zero to Extrapolated Infinite Time [MRAUC(0-∞)]
Description: Molar ratio of metabolite to parent area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞) [MRAUC(0-∞)].
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
Ratio | 0.1371 (0.0188) | 0.2239 (0.0398)

14. Secondary Outcome: Metabolite to Parent Ratio of Maximum Observed Plasma Concentration (MRCmax)
Description: Metabolite to parent molar ratio of maximum observed plasma concentration (Cmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Number analyzed (Participants) | 15 | 15
Ratio | 0.2469 (0.0634) | 0.2766 (0.0511)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Crizotinib 150 mg | Crizotinib 150 mg + Ketoconazole 200 mg BID
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib 150 mg (N=15) | Crizotinib 150 mg + Ketoconazole 200 mg BID (N=15)
Abnormal sensation in eye (Eye disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Nodule (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.